CLINICAL TRIAL: NCT05725278
Title: Health Impact Evaluation of Triggerise's Tiko Platform
Brief Title: Impact Evaluation of Triggerise's Tiko Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Network for Engineering and Economics Research and Management (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Triggerise Protocol V2
Record Dates: First submitted 2023-01-12; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Contraception; Iron Deficiency Anemia of Pregnancy; Antenatal Care; Postnatal Care
Keywords: mHealth; Social Franchising; Social Marketing; Impact Evaluation; Market-Driven; Family Planning; Antenatal Care; Community Health Workers
MeSH Terms: interventions — Standard of Care; Commerce

STUDY DESIGN:
Intervention Model Description: The study compares family planning, antenatal care and postnatal care related outcomes (multiple) for women who had registered on Tiko Platform between those who used the platform and those who did not access any services on the platform. The comparison is done ex-post with a single cross sectional survey in March-April 2021. Model uses fixed effects at Pro-Agent level who is a local health promoter of a small geographical area and recruits and serves women in that area so that confounders at agent and levels beyond are controlled. For women/household level confounder control, a few socio-economic and demographic variables at the woman level were included in the model, and sensitivity of the results with and without adjusting for these control variables was investigated.
Masking Description: By nature of the intervention, the implementers or pro agents knew who the users and non-users are, and this was critical even in sampling. The data collectors did not know who were the users and non-users but a smart data collector / outcome assessor could figure out who were the users based on type of questions that were asked and answered. Investigators also knew who were users and non users as it was essential for analysis and setting up the data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Users of Tiko Platform (Experimental): These participants accessed various services on Tiko platform such as buying contraceptives, visiting doctors for ANC etc. They earned Tiko Miles/Points for such health seeking behaviours which they could then redeem at network of grocery shops, pharmacies, beauty salon etc. Tiko card also enabled them to get discounts at pharmacies and at health care providers. These participants were free to access any other government or private health care facility as free economic agents. Users of Tiko platform were identified by the backend system that recorded all health seeking behaviours / actions, reward point accumulation, and use of those reward points.
  Interventions: Behavioral: Tiko Platform Behavioural cum mHealth Intervention
- Non-Users of Tiko Platform (Active Comparator): These participants registered on Tiko platform on basis of recruitment drive and pitch by Pro agents, but they did not access any service and became dormant. However, These participants were free to access any other government or private health care facility and could access fame family planning and ANC products and services. They could even access Tiko network doctors and pharmacies but they would not get any Tiko Miles/Points or discounts without the use of Tiko card. Non Users were identified as those registered women who did not have any record of using services using Tiko card as per the backend system
  Interventions: Other: Standard of Care / Business as Usual

INTERVENTIONS:
Behavioral: Tiko Platform Behavioural cum mHealth Intervention — Tiko platform is a mix of social franchising and social marketing concepts to promote health behaviours through rewards to health promoters (pro agents), healthcare providers (doctors and pharmacies), Beneficiaries (women needing FP and/or ANC services), and shop keepers and life-style service providers where beneficiaries, providers and promoters could use their rewards points. The health promoters could purchase from wholesale retailers products such as sanitary napkins, condoms and then resale these at profit. Beneficiaries were given discounts and their rewards points can be used as cash to avail certain lifestyle services at participating locations, and so did the health care providers. Pro agents also got incentives for recruiting the beneficiaries and after beneficiaries reached certain service access/use milestones. All this was integrated on a mHealth platform using smart phones and smart cards (for those without access to Tiko card).
  Arms: Users of Tiko Platform
Other: Standard of Care / Business as Usual — Non-Users of Tiko did not use Tiko platform but they could access any health care provider or pharmacy to avail same services related to Family planning, antenatal care, postnatal care
  Arms: Non-Users of Tiko Platform

SUMMARY:
Triggerise designed web and phone based Tiko platform to connect young girls and women to the health products, services and information. The platform uses principles of behaviour economics to motivate positive choices-including rewards, promotions, discounts, coupons, reminders, alerts etc. The platform was implemented in several cities from seven states of India to provide Sexual Reproductive Health (SRH) and maternal and child health (MCH) products and services. The consumers (called Rafikis) use Tiko card to get discounts and to earn 'Tiko miles' rewards at Tiko franchised healthcare providers and pharmacies. Tiko miles are redeemable towards lifestyle products or services (e.g., beauty salons). The local Tiko health promoter (celled Pro agent) can also buy health and hygiene products at bulk discounts and sell them at profit.

Triggerise appointed Network for Engineering, Economics Research and Management (NEERMAN) to conduct an independent impact assessment of the Tiko platform with multiple research objectives include health impact evaluation at the Rafiki level.

NEERMAN used an ex-post observational design to compare usage of SRH and MCH services and family planning (FP), antenatal care (ANC) and postnatal care (PNC) practices by comparing Users and Non-Users of Tiko platform, and accounting for the selection bias statistically. The structured questionnaire collected data on knowledge, practices, barriers, enablers for SRH and MCH services, exposure o Tiko platform, and how it helped or did not help. The survey participants were approx. 1200 users and 600 non-users being served by approx. 350 pro-agents in their respective operations area.

The association between use of Tiko platform and various outcomes were identified using a generalized linear model with fixed effects at pro-agent level and including a set of covariates. To evaluate the effect modification by type of pro agent - government community health worker (CHW) versus others - an interaction model was used. The standard errors were automatically clustered at pro-agent level due to fixed effects. Primary outcomes are proportion of married Rafikis currently using any contraceptives, currently using modern short-term contraceptives, proportion of Rafikis who delivered a child post Jan 2019 and received at least 4 ANC check-ups, consumed at least 100 iron folic acid (IFA( during pregnancy, and received a PNC check-up within 6 weeks of birth.

DETAILED DESCRIPTION:
See subsequent sections

ELIGIBILITY:
Inclusion Criteria:

* Women who are registered on Tiko Platform with Pro-agents active in 2020-21
* Age 18-50
* Address and contacts details are found with help of Pro-agent

Exclusion Criteria:

* Does not consent to participation
* Does not agree or confirm registering on Tiko Platform
* If a woman is never married, she is excluded from survey on family planning but surveyed for use of Tiko platform
* If a married woman does not have a child born on/after 1 January 2019, then she is excluded from the survey on antenatal care, delivery and postnatal care but surveyed for use of Tiko platform

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1708 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Proportion of women currently using any contraceptives | Through survey completion, an average of 1 month
  Whether a woman used any contraceptive - traditional or modern methods, and permanent or temporary methods
Proportion of women currently using modern short-term contraceptives | Through survey completion, an average of 1 month
  Whether a woman used modern and temporary contraception methods
Proportion of women who consumed 100 or more Iron Folic Acid (IFA) tablets during last pregnancy | 9 months during pregnancy with the youngest child
  Whether the study participant recalled consuming 100 or more IFA tablets when pregnant with youngest child born after 1 January 2019
Proportion of women who received 4 or more antenatal check-ups during last pregnancy | 9 months during pregnancy with the youngest child
  Whether the study participant recalled receiving 4 or more ANC check-ups from any health care provider when pregnant with youngest child born after 1 January 2019
Proportion of women who received a postnatal check-up within 6 week of the delivery from a healthcare provider | Within 6 weeks after delivery of the youngest child
  Whether the study participant recalled receiving at least one postnatal health check up within 6 weeks of the youngest child's birth

SECONDARY OUTCOMES:
Out of pocket expenditure on antenatal care, iron folic acid tablets, delivery, and postnatal check-ups | 9 months during pregnancy with the youngest child
  Reported expenditure in Indian Rupees for antenatal care, iron folic acid tablets, delivery, and postnatal check-ups associated with the youngest child born after 1 January 2019
Out of pocket expenditure on Family planning services and products | Past 24 months (from survey date)
  Reported expenditure in Indian Rupees for permanent or temporary contraceptive methods
Proportion of women receiving Antenatal check-ups at (a) Tiko franchisee doctors, (b) other private doctors, or (c) government healthcare provider | 9 months during pregnancy with the youngest child
  Separate proportions are estimated for each of the three locations of antenatal check-ups when pregnant with youngest child born after 1 January 2019
Proportion of women receiving postnatal check-ups at (a) Tiko franchisee doctors, (b) other private doctors, or (c) government healthcare provider | Within 6 weeks after delivery of the youngest child
  Separate proportions are estimated for each of the three locations of postnatal check-ups within 6 weeks after delivery of the youngest child born after 1 January 2019

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Patil, PhD, Principal Investigator — Network for Engineering and Economics Research and Management
Locations (1):
- NEERMAN, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No
While NEERMAN holds data use and publication rights from Triggerise, the data ownership rests with Triggerise so data access to de-identify observations and variables used in pit is unclear published papers can be made available under certain conditions

REFERENCES:
- [Derived] Patil SR, Gopalakrishnan L, Sai VS, Matikanya R, Rajpal P. Markets, incentives, and health promotion can improve family planning and maternal health practices: a quasi-experimental evaluation of a tech-enabled social franchising and social marketing platform in India. BMC Public Health. 2024 Jan 23;24(1):264. doi: 10.1186/s12889-023-17413-w. PMID 38262982

DOCUMENTS (2):
  • Study Protocol (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT05725278/Prot_000.pdf
  • Informed Consent Form (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/78/NCT05725278/ICF_001.pdf